CLINICAL TRIAL: NCT05038475
Title: Longitudinal Observation of Clinical and Immunological Profiles After SARS-Cov-2 Infection
Brief Title: Clinical and Immunological Responses After SARS-CoV-2 Infection Causing COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Association "Naso Sano" Onlus (Other)
Responsible Party: Principal Investigator, Dr. Puya Dehgani Mobaraki, Principal Investigator, Association "Naso Sano" Onlus
Other Study IDs: ANS-2020/001
Record Dates: First submitted 2021-06-10; First posted 2021-09-09 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Covid19; SARS-CoV2 Infection; Olfactory Disorder; COVID-19; Smell Loss; Smell Disorder
Keywords: Antibody responses; olfaction; smell; sars-cov-2; covid-19; IgG; IgM; serology; immune response; humoral response
MeSH Terms: conditions — COVID-19; Anosmia; Olfaction Disorders | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild group: As per the WHO guidelines, the patients were divided into two groups based on disease severity: Mild and Moderately severe.
  This was based on the self-reported symptoms experienced by the patients during the infection period (March 2020).
  Intervention:
  COVID-19 Antibody testing at different time points
  Interventions: Diagnostic Test: COVID-19 antibody test
- Moderately-severe group: As per the WHO guidelines, the patients were divided into two groups based on disease severity: Mild and Moderately severe.
  This was based on the self-reported symptoms experienced by the patients during the infection period (March 2020).
  Intervention:
  COVID-19 Antibody testing at different time points
  Interventions: Diagnostic Test: COVID-19 antibody test

INTERVENTIONS:
Diagnostic Test: COVID-19 antibody test — FDA-approved Immunoassays were used in the study. At the beginning of the study, up to 3 months, ELISA and CLIA immunoassays were adopted to analyze the antibody titers. Thereafter, CLIA was used for longitudinal analysis of antibody titers for consecutive months. Anti

SUMMARY:
There are very few long-term studies that analyze the immune responses in patients recovered from COVID-19 caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

The main aim of this study is to analyze the clinical profile and immune responses of recovered COVID-19 patients in a representative cohort of people in the Umbria region of Italy. The participants had a history of testing positive for SARS-CoV-2 in March 2020 by Reverse Transcriptase- Quantitative Polymerase Chain Reaction (RT-qPCR). The participants were invited for voluntary participation in a seroprevalence study. This study analyzes longitudinally the presence of antibodies against SARS-CoV-2 by sequential serological tests at different time points using two FDA-approved Immunoassays. At the first serum sample collection, the participants were asked to provide information about their COVID-19 clinical history including clinical profile, co-morbidities, and treatment undertaken using a standardized questionnaire. Successive sequential serological assessments were conducted to understand the immune responses in these recovered patients.

Moreover, stage two of the study involves, analysis of antibody titers in recovered vaccinated individuals and their follow-up.

DETAILED DESCRIPTION:
Study design: A monocentric pilot longitudinal observational study

Study subjects: patients recovered from SARS-CoV-2 infection in March 2020 (detected by RT-PCR)

Study method: The study was conducted after written informed consent for voluntary participation. The antibody titers were longitudinally analyzed by sequential serological tests at different time points (TPs) using two FDA-approved Immunoassays. At the first serum sample collection, the participants were asked to provide information about their COVID-19 clinical history including clinical profile, co-morbidities, and the treatment undertaken using a standardized questionnaire.

From May 2020 to January 2021:

Anti-Nucleocapsid (NCP) antibodies were analyzed using FDA-approved CLIA immunoassay through sequential serum samples.

Time was treated as a factor and six different time points (TPs) were defined (T0-T5). The first blood sample was collected in the month of May 2020, 2 months after the month of infection (March), and was defined as T0. Consecutive serological samples were analyzed at different TPs; three months (T1), five months (T2), seven months (T3), eight months (T4), and ten months (T5) post-infection in June, August, October, November of 2020 and January 2021 respectively.

At this point, a more specific immunoassay was adopted to detect neutralizing antibodies against the Spike-Receptor binding domain for future assessments.

From late February 2021:

an additional n=12 patients (8 female and 4 male), who met the eligibility criteria for participation, were enrolled in the study and added to the original cohort (n=30). These patients (n=12), similar to the original cohort, had a history of testing positive for SARS-CoV-2 by RT-qPCR in March 2020, updating the sample size to n=42.

Since the legal provisions adopted by the Italian Ministry of Health advised mandatory vaccination for all Healthcare Workers, irrespective of previous disease status, n=10 patients (4 female and 6 male) were gradually vaccinated from mid-March 2021 and hence excluded from the original cohort, making the revised final sample size as n=32.

The presence of antibodies was analyzed The study continues to actively enroll patients for future analysis.

with vaccination in progress, the antibody titers of the recovered and then vaccinated patients will also be analysed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who tested positive for SARS-CoV-2 in March 2020. These patients will be divided into two groups and followed up over time. The first group will include patients who have recovered and have not received the vaccine. The second group will include patients who have recovered and have received the vaccine.
2. No acute respiratory infection or active SARS-CoV-2 infection.
3. Informed consent of the adult participant.

Exclusion Criteria:

1. Individuals <18 years or >80 years.
2. No informed consent by the adult participant.
3. Suspicion of acute COVID-19 infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who tested positive for SARS-CoV-2 in March 2020 and are not vaccinated till date, within the age range of 18-80 years, with no active respiratory infection / active COVID-19 infection and willing to give informed consent were invited to take part in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Analysis of demographic profile (Age) of recovered COVID-19 patients [at inclusion] | At inclusion
  Demographic profile included Age at presentation (in years)
Analysis of demographic profile (Gender) of recovered COVID-19 patients [at inclusion] | At inclusion
  Demographic profile included Sex (gender) at presentation (male/female/other)
Analysis of demographic profile (occupation) of recovered COVID-19 patients [at inclusion] | At inclusion
  Demographic profile included occupation at presentation (healthcare-worker/non-healthcare)
Analysis of clinical profile of recovered COVID-19 patients [at inclusion] | At inclusion
  Clinical profile included clinical symptoms experienced at the time of presentation. The participant completed a questionnaire with "Yes" or "no" for each symptom. The symptoms were namely: Fever, Rhinorrhea, Dry cough, Sore throat, Shortness of breath, fatigue, Headche, Muscle ache, skin eruptions, diarrhoea, conjunctivitis, loss of smell, loss of taste, chest pain or any other symptom (please specify).
Analysis of associated co-morbidities in recovered COVID-19 patients [at inclusion] | At inclusion
  Participants completed a questionnaire with "Yes" or "no" for history of comorbidities namely: Asthma/seasonal allergies, Diabetes Mellitus, Hypertension, cardiovascular disease or any other co-morbidity (please specify).
Analysis of immunological profile recovered COVID-19 patients [at inclusion] | At inclusion
  The participants were questioned about their respective blood groups.
Seroprevalence of IgM and IgG against Nucleocapsid of SARS-CoV-2 (in AU/ml) [from T0 to T5] | 8 months
  From May 2020 to January 2021, anti-nucleocapsid (NCP) antibodies developed against SARS-CoV-2 were analysed using n-CoV IgM/IgG CLIA assay through sequential serological tests in n=30 patients. Time was treated as a factor and six time points were defined. The first blood sample was collected in May 2020 (2 months after infection) and was defined as T0. Consecutive samples were analysed at 3 months (T1), five months (T2) , seven months (T3) and eight months (T4) and ten months (T5) post infection in June, August, October, November of 2020 and January 2021 respectively.
Seroprevalence of IgM and IgG against spike-receptor binding domain of SARS-CoV-2 (in AU/ml) [from T6 to T8] | through study completion, an average of 2 years
  A more specific immunoassay (CLIA) against SARS-CoV-2 S-RBD was adopted for future assessments. From late February 2021, an additional n = 12 patients (8 female and 4 male), who met the eligibility criteria for participation, were enrolled in the study and added to the original cohort (n = 30). These patients (n=12), similar to the original cohort, had a history of testing positive for SARS-CoV-2 by RT-qPCR in March 2020, updating the sample size to n = 42. Since the legal provisions adopted by the Italian Ministry of Health advised mandatory vaccination for all Healthcare Workers, irrespective of previous disease status,n=10 patients (4 female, 6 male) were gradually vaccinated from mid-March 2021 and excluded from the original cohort, making the revised final sample size,n = 32.
Seroprevalence of IgM and IgG against spike-receptor binding domain of SARS-CoV-2 (in AU/ml) for vaccinated individuals | through study completion, an average of 2 years
  The vaccinated recovered individuals continued to report for follow-up for antibody analysis

SECONDARY OUTCOMES:
Co-relation of demographic profile with antibody titers against NCP of SARS-CoV-2 with respect to disease severity [ Time Frame: at inclusion and within observational period ] | 8 months
  Demographic profile such as Age, Sex, occupation were analysed to look for any association with disease severity and antibody titers against NCP at different time points from (T0-T5)
Co-relation of demographic profile with antibody titers against spike- RBD of SARS-CoV-2 with respect to disease severity [ Time Frame: at inclusion and within observational period ] | 4 months
  Demographic profile such as Age, Sex, occupation were analysed to look for any association with disease severity and antibody titers against spike-RBD at different time points from (T6-T8)
Co-relation of symptoms and antibody titer levels against Nucleocapsid of SARS-CoV-2 with respect to disease severity [ Time Frame: at inclusion and within observational period ] | at inclusion and within the observational period (8 months)
  Presence of symptoms (in March 2020) suggestive of a common cold, influenza and similar upper respiratory tract infections with help of questionnaire.
  Symptoms recorded : Fever , Rhinorrea, Dry cough, sore throat, Shortness of breath, Headache, skin eruptions, muscle ache, diarrhoea, conjunctivitis, loss of smell, loss of taste, chest pain and its association with disease severity and antibody titers against NCP at different time points (T0-T5).
Co-relation of self reported symptoms and antibody titer levels against spike-RBD with respect to disease severity [ Time Frame: at inclusion and within observational period ] | at inclusion and within the observational period (4 months)
  Presence of symptoms (in March 2020) suggestive of a common cold, influenza and similar upper respiratory tract infections with help of questionnaire.
  Symptoms recorded : Fever , Rhinorrea, Dry cough, sore throat, Shortness of breath, Headache, skin eruptions, muscle ache, diarrhoea, conjunctivitis, loss of smell, loss of taste, chest pain and its association with antibody titers against spike receptor binding domain with respect to disease severity at different time points (T6-T8).
Co-relation of co-morbidities and antibody titer levels with respect to disease severity [ at inclusion] | at inclusion and within the observational period (8 months)
  history of asthma/ allergies/diabetes/hypertension/cardiovascular diseases and its association with disease severity and anti-NCP antibody titers (quantitative) at different time points (T0-T5)
Co-relation of co-morbidities and antibody titer levels with respect to disease severity [ at inclusion] | at inclusion and within the observational period (through study completion, an average of 2 years)
  history of asthma/ allergies/diabetes/hypertension/cardiovascular diseases and its association with disease severity and anti-S-RBD antibody titers (quantitative) at different time points (T6-T8)
Co-relation of antibody titer levels and smell and taste dysfuntion with respect to disease severity [ at inclusion] | at inclusion and within the observational period (through study completion, an average of 2 years)
  history of asthma/ allergies/diabetes/hypertension/cardiovascular diseases and its association with disease severity and anti-S-RBD antibody titers (quantitative) at different time points (T6-T8)

CONTACTS AND LOCATIONS:
Overall Officials: Puya Dehgani-Mobaraki, MD, Principal Investigator — Associazione Naso sano, Italy
Locations (1):
- Associazione Naso Sano, San Mariano, Perugia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Sensitive clinical data from the patients will be collected. Therefore, it is not yet decided, if it will be possible to share IPD while preserving participant anonymity and privacy.

REFERENCES:
- [Result] Abu-Raddad LJ, Chemaitelly H, Coyle P, Malek JA, Ahmed AA, Mohamoud YA, Younuskunju S, Ayoub HH, Al Kanaani Z, Al Kuwari E, Butt AA, Jeremijenko A, Kaleeckal AH, Latif AN, Shaik RM, Abdul Rahim HF, Nasrallah GK, Yassine HM, Al Kuwari MG, Al Romaihi HE, Al-Thani MH, Al Khal A, Bertollini R. SARS-CoV-2 antibody-positivity protects against reinfection for at least seven months with 95% efficacy. EClinicalMedicine. 2021 May;35:100861. doi: 10.1016/j.eclinm.2021.100861. Epub 2021 Apr 28. PMID 33937733
- [Result] Piccoli L, Park YJ, Tortorici MA, Czudnochowski N, Walls AC, Beltramello M, Silacci-Fregni C, Pinto D, Rosen LE, Bowen JE, Acton OJ, Jaconi S, Guarino B, Minola A, Zatta F, Sprugasci N, Bassi J, Peter A, De Marco A, Nix JC, Mele F, Jovic S, Rodriguez BF, Gupta SV, Jin F, Piumatti G, Lo Presti G, Pellanda AF, Biggiogero M, Tarkowski M, Pizzuto MS, Cameroni E, Havenar-Daughton C, Smithey M, Hong D, Lepori V, Albanese E, Ceschi A, Bernasconi E, Elzi L, Ferrari P, Garzoni C, Riva A, Snell G, Sallusto F, Fink K, Virgin HW, Lanzavecchia A, Corti D, Veesler D. Mapping Neutralizing and Immunodominant Sites on the SARS-CoV-2 Spike Receptor-Binding Domain by Structure-Guided High-Resolution Serology. Cell. 2020 Nov 12;183(4):1024-1042.e21. doi: 10.1016/j.cell.2020.09.037. Epub 2020 Sep 16. PMID 32991844
- [Result] Suthar MS, Zimmerman MG, Kauffman RC, Mantus G, Linderman SL, Hudson WH, Vanderheiden A, Nyhoff L, Davis CW, Adekunle O, Affer M, Sherman M, Reynolds S, Verkerke HP, Alter DN, Guarner J, Bryksin J, Horwath MC, Arthur CM, Saakadze N, Smith GH, Edupuganti S, Scherer EM, Hellmeister K, Cheng A, Morales JA, Neish AS, Stowell SR, Frank F, Ortlund E, Anderson EJ, Menachery VD, Rouphael N, Mehta AK, Stephens DS, Ahmed R, Roback JD, Wrammert J. Rapid Generation of Neutralizing Antibody Responses in COVID-19 Patients. Cell Rep Med. 2020 Jun 23;1(3):100040. doi: 10.1016/j.xcrm.2020.100040. Epub 2020 Jun 8. PMID 32835303
- [Result] Sette A, Crotty S. Adaptive immunity to SARS-CoV-2 and COVID-19. Cell. 2021 Feb 18;184(4):861-880. doi: 10.1016/j.cell.2021.01.007. Epub 2021 Jan 12. PMID 33497610